CLINICAL TRIAL: NCT02771977
Title: Drug-Targeted Alerts for Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000025786; 1R01DK113191-01A1 (NIH)
Record Dates: First submitted 2016-05-11; First posted 2016-05-13 (Estimated); Results first posted 2023-06-29 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): No alert will be fired.
- Drug-specific alert (Experimental): A drug-specific AKI alert, including information about the drug of interest as well as the presence of AKI will be fired.
  Interventions: Other: Drug-specific alert

INTERVENTIONS:
Other: Drug-specific alert — A drug-specific alert, informing the provider of the presence of AKI as well as recent exposure to a potentially nephrotoxic agent, will be fired.
  Arms: Drug-specific alert

SUMMARY:
In this trial, patients with acute kidney injury who have recently received a drug that may affect kidney function will be randomized to having an alert placed in the electronic health record or usual care.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) carries a significant, independent risk of mortality among hospitalized patients. Recent studies have demonstrated increased mortality among patients with even small increases in serum creatinine concentration. International guidelines for the treatment of AKI focus on appropriate management of drug dosing, avoiding nephrotoxic exposures, and careful attention to fluid and electrolyte balance. Early nephrologist involvement may also improve outcomes in AKI. Without appropriate provider recognition of AKI, however, none of these measures can be taken, and patient outcomes may suffer. AKI is frequently overlooked by clinicians, but carries a substantial cost, morbidity and mortality burden.

Our research group recently conducted a large-scale multicenter randomized controlled trial of electronic alerts for AKI throughout the Yale New Haven Health System from 2018 to 2020. The trial, which enrolled 6,030 patients with AKI, randomized patients between usual care and an intervention group whereby providers received a general AKI alert informing them to the presence of AKI and the patient's recent creatinine trends, and provided a link to an AKI-specific order set. Our study showed that, overall, alerting physicians to the presence of AKI did not demonstrate a difference in the rate of our primary outcome of progression of AKI, dialysis, or death, nor were there any differences in process measures accessed (i.e. provider actions) between the two groups, however, there was substantial heterogeneity among the study sites. Given the highly heterogenous nature of AKI, a more personalized approach may be warranted. Further, this study enrolled all patients who developed AKI rather than a targeted subset of patients who may benefit, such as those AKI patients receiving potentially harmful kidney-toxic medications. In the present proposal, we seek to expand upon our prior study to determine if the use of medication targeted electronic alerts will modify provider behavior, particularly in regards to nephrotoxic medication use and cessation, in the care of hospitalized patients with AKI and/or reduce the rates of progression to AKI, dialysis, or mortality in hospitalized patients.

The current study is a randomized, controlled trial of a medication-targeted electronic AKI alert system. Using the Kidney Disease: Improving Global Outcomes (KDIGO) creatinine criteria, inpatients at 4 different teaching hospitals of the Yale New Haven Health System that have had at least one dose of a nephrotoxic agent of interest within 24 hours of AKI onset will be randomized to either usual care or a medication-targeted alert that informs the provider of the presence of AKI and the patient's recent exposures to the targeted classes of medications with an option to discontinue. The primary outcome will be a composite of AKI progression, dialysis, or mortality within 14 days of randomization. Secondary outcomes will focus on the rate of cessation of any medication of interest within 24 hours of randomization and various other best practice metrics.

ELIGIBILITY:
Inclusion Criteria:

* Acute Kidney Injury based upon the Kidney Disease: Improving Global Outcomes creatinine criteria (a 0.3mg/dl increase over 48 hours or 50% increase over 7 days) and an active order within the past 24 hours to one of the following classes of medications:
* Non-steroidal anti-inflammatory drug
* Renin Angiotensin Aldosterone System Antagonists
* Proton Pump Inhibitors

Exclusion Criteria:

* Dialysis order prior to AKI onset
* Previous randomization
* Admission to a hospice service or CMO
* First hospital creatinine >=4.0 mg/dl
* ESKD diagnosis code
* Kidney transplant within six months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5060 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Wissel BD, Percy Z, Zachem TJ, Beaulieu-Jones B, Kohane IS, Goldstein SL, Gecili E, Dexheimer JW. Heterogenous effect of automated alerts on mortality. J Am Med Inform Assoc. 2025 Dec 25:ocaf222. doi: 10.1093/jamia/ocaf222. Online ahead of print. PMID 41445428
- [Derived] Wissel BD, Percy Z, Zachem TJ, Beaulieu-Jones B, Kohane IS, Goldstein SL, Gecili E, Dexheimer JW. Heterogeneous Effect of Automated Alerts on Mortality. medRxiv [Preprint]. 2025 Aug 13:2025.08.11.25333302. doi: 10.1101/2025.08.11.25333302. PMID 40832403
- [Derived] Wilson FP, Yamamoto Y, Martin M, Coronel-Moreno C, Li F, Cheng C, Aklilu A, Ghazi L, Greenberg JH, Latham S, Melchinger H, Mansour SG, Moledina DG, Parikh CR, Partridge C, Testani JM, Ugwuowo U. A randomized clinical trial assessing the effect of automated medication-targeted alerts on acute kidney injury outcomes. Nat Commun. 2023 May 17;14(1):2826. doi: 10.1038/s41467-023-38532-3. PMID 37198160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and enrollment was done automatically via our best practice alert, which analyzed hospitalized patients for inclusion and exclusion criteria and, if met, automatically enrolled and randomized patients to the usual care or alert group.
Pre-assignment Details: 5,839 subjects were assessed for eligibility, with 779 excluded due to either the patient's admission dates being prior to the alert becoming active, the first alert firing after a discharge order, or because the patient was already randomized in a previous hospital admission. 5,060 patients were then randomized to alert versus usual care with zero loss to follow up.
Period: Overall Study
Arm/Group | Usual Care | Drug-specific Alert
Started | 2528 | 2532
Completed | 2528 | 2532
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Drug-specific Alert | Total
Number analyzed (Participants) | 2528 | 2532 | 5060
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 70 [59 to 80] | 70 [59 to 81] | 70 [59 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1222 | 1231 | 2453
  Male | 1306 | 1301 | 2607
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 341 | 350 | 691
  Not Hispanic or Latino | 2163 | 2166 | 4329
  Unknown or Not Reported | 24 | 16 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 11 | 18
  Asian | 40 | 40 | 80
  Native Hawaiian or Other Pacific Islander | 1 | 5 | 6
  Black or African American | 470 | 498 | 968
  White | 1714 | 1683 | 3397
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 296 | 295 | 591
Hospital Location [Count of Participants; unit: Participants]
  Medical Admission | 1924 | 1937 | 3861
  ICU | 598 | 560 | 1158
  Emergency Department | 87 | 90 | 177
  Ward | 1746 | 1775 | 3521
Hospital [Count of Participants; unit: Participants]
  Hospital 1 | 1250 | 1197 | 2447
  Hospital 2 | 591 | 623 | 1214
  Hospital 3 | 446 | 464 | 910
  Hospital 4 | 241 | 248 | 489
Comorbidities [Count of Participants; unit: Participants]
  Chronic Kidney Disease | 616 | 671 | 1287
  Congestive Heart Failure | 784 | 827 | 1611
  Chronic Obstructive Pulmonary Disorder (COPD) | 762 | 776 | 1538
  Diabetes Mellitus | 928 | 967 | 1895
  Hypertension | 1726 | 1710 | 3436
  Malignancy | 563 | 549 | 1112
  Depression | 580 | 601 | 1181
  Liver Disease | 359 | 310 | 669
Acute Kidney Injury (AKI) stage at randomization [Count of Participants; unit: Participants] — Stages of Acute Kidney Injury (AKI) were defined using the Kidney Disease Improving Global Outcomes (KDIGO) serum creatinine (SCr) criteria, with increasing stages representing more progressive disease:
  Stage 1: An increase in SCr by greater than or equal to 0.3 mg/dL within 48 hours; or an increase in SCr by greater than or equal to 1.5 times baseline within 7 days Stage 2: An increase in SCr by 2.0 to 2.9 times baseline Stage 3: An increase in SCr by 3.0 times baseline or greater Stage 0: Randomized patients without AKI due to lab error
  Participants
    Stage 0 | 3 | 6 | 9
    Stage 1 | 2248 | 2279 | 4527
    Stage 2 | 230 | 191 | 421
    Stage 3 | 47 | 56 | 103
Estimated Glomerular Filtration Rate (eGFR) on admission [Median (Inter-Quartile Range); unit: ml/min/1.73m^2] | 61 [38 to 88] | 60 [38 to 87] | 60.3 [38.5 to 87.5]
Creatinine at randomization [Median (Inter-Quartile Range); unit: mg/dL] | 1.5 [1.1 to 2] | 1.5 [1.2 to 2] | 1.5 [1.2 to 2]
Creatinine at admission [Median (Inter-Quartile Range); unit: mg/dL] | 1.2 [0.8 to 1.6] | 1.2 [0.9 to 1.7] | 1.2 [0.8 to 1.6]
Sodium [Median (Inter-Quartile Range); unit: meq/L] | 138 [135 to 141] | 138 [135 to 141] | 138 [135 to 141]
Potassium [Median (Inter-Quartile Range); unit: meq/L] | 4.2 [3.8 to 4.6] | 4.2 [3.8 to 4.6] | 4.2 [3.8 to 4.6]
Chloride [Median (Inter-Quartile Range); unit: meq/L] | 102 [99 to 106] | 102 [99 to 106] | 102 [99 to 106]
Bicarbonate [Median (Inter-Quartile Range); unit: meq/L] | 23 [20 to 26] | 23 [21 to 26] | 23 [20 to 26]
Anion gap [Median (Inter-Quartile Range); unit: meq/L] | 12 [10 to 14] | 12 [10 to 14] | 12 [10 to 14]
Blood urea nitrogen (BUN) [Median (Inter-Quartile Range); unit: mg/dL] | 29 [19 to 42] | 29 [20 to 42] | 29 [19 to 42]
White blood cell count [Median (Inter-Quartile Range); unit: x1000/uL] | 9.6 [6.7 to 13.6] | 9.5 [6.8 to 13.5] | 9.6 [6.7 to 13.6]
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 10.6 [8.9 to 12.4] | 10.6 [8.8 to 12.5] | 10.6 [8.8 to 12.5]
Platelet count [Median (Inter-Quartile Range); unit: x1000/uL] | 214 [149 to 288] | 213 [153 to 287] | 213 [151 to 288]
Modified SOFA score [Median (Inter-Quartile Range); unit: Scores on a scale] — The Modified Sequential Organ Failure Assessment (SOFA) score assesses the performance of several organ systems and helps predict ICU mortality. There are six distinct scores that make up the SOFA score (respiratory, cardiovascular, hepatic, coagulation, renal, and neurological) that can range from 0 (normal) to 4 (most abnormal), with a minimum total SOFA score of 0 and a maximum SOFA score of 24. A higher score indicates a greater risk of mortality.
  Scores on a scale | 3 [1 to 5] | 2 [1 to 4] | 2 [1 to 4]
Exposures prior to AKI [Count of Participants; unit: Participants]
  Contrast in prior 72 hours | 662 | 621 | 1283
  Renin angiotensin aldosterone system inhibitors (RAASi) | 1329 | 1350 | 2679
  (Non-steroidal anti-inflammatory drugs (NSAIDs) | 805 | 748 | 1553
  (Proton pump inhibitors (PPIs) | 1644 | 1654 | 3298
  Patients on one medication of interest (RAASi, NSAID, or PPI) | 1451 | 1470 | 2921
  Patients on two medications of interest (RAASi, NSAID, or PPI) | 904 | 904 | 1808
  Patients on three medications of interest (RAASi, NSAID, or PPI) | 173 | 158 | 331

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Progression of AKI OR Dialysis OR Death
Description: Progression of AKI is defined by an increase in KDIGO creatinine stage from time of randomization to the present. Dialysis is defined by the receipt of hemodialysis, continuous renal replacement therapy or peritoneal dialysis. Isolated ultrafiltration treatments will not be included. Mortality will be determined from hospital records.
Time Frame: 14 days from Randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Drug-specific Alert
Number analyzed (Participants) | 2528 | 2532
Participants | 639 | 585

2. Secondary Outcome: Percentage of Patients for Whom Any One of the Targeted Medications is Discontinued
Description: The Percentage of patients for whom the targeted agent was discontinued within 24 hours from randomization. For individuals with active orders for more than one targeted agent, cessation of any will be adequate to meet this endpoint.
Time Frame: Assessed within 24 hours from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Drug-specific Alert
Number analyzed (Participants) | 2528 | 2532
Participants | 1413 | 1547

3. Secondary Outcome: 14- Day Mortality Rate
Description: Percentage of patients who expire within 14 days of randomization
Time Frame: Assessed from date of randomization to date of death from any cause, within 14 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Drug-specific Alert
Number analyzed (Participants) | 2528 | 2532
Participants | 282 | 253

4. Secondary Outcome: Inpatient Mortality Rate
Description: Percentage of patients who expire during index hospitalization.
Time Frame: Assessed from point of randomization to the date of death from any cause during the end of current index hospitalization, up to 365 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Drug-specific Alert
Number analyzed (Participants) | 2528 | 2532
Participants | 365 | 356

5. Secondary Outcome: Percentage of Patients Who Receive Dialysis Within 14 Days of Randomization
Description: Receipt of hemodialysis, continuous renal replacement, or peritoneal dialysis within 14 days of randomization
Time Frame: Assessed from point of randomization to date of first documented dialysis order, within 14 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Drug-specific Alert
Number analyzed (Participants) | 2528 | 2532
Participants | 127 | 123

6. Secondary Outcome: Percentage of Patients on Inpatient Dialysis
Description: Receipt of hemodialysis, continuous renal replacement, or peritoneal dialysis during index hospitalization
Time Frame: Assessed from point of randomization to the date of first documented dialysis order during index hospitalization, up to 365 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Drug-specific Alert
Number analyzed (Participants) | 2528 | 2532
Participants | 137 | 151

7. Secondary Outcome: Percentage of Patients Discharged on Dialysis
Description: Active orders for dialysis at the point of discharge from the index hospitalization
Time Frame: Assessed at the point of discharge from index hospitalization, up to 365 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Drug-specific Alert
Number analyzed (Participants) | 2528 | 2532
Participants | 105 | 127

8. Secondary Outcome: Percentage of Patients With AKI Progression From Stage 1 to Stage 2
Description: Progression to stage 2 AKI, represented by a doubling of baseline creatinine levels.
Time Frame: Assessed from date of randomization to date of documented AKI progression, within 14 days of randomization
Population: Population analyzed represents the number of subjects with AKI Stage 1 upon enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Drug-specific Alert
Number analyzed (Participants) | 2248 | 2279
Participants | 248 | 242

9. Secondary Outcome: Percentage of Patients With AKI Progression From Stage 2 to Stage 3
Description: Progression to stage 3 AKI, represented by a tripling of baseline creatinine levels.
Time Frame: Assessed from date of randomization to date of documented AKI progression, within 14 days of randomization
Population: Analyzed population includes subjects with Stage 1 or Stage 2 AKI upon enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Drug-specific Alert
Number analyzed (Participants) | 2478 | 2470
Participants | 256 | 231

10. Secondary Outcome: AKI Duration
Description: Time in hours between AKI onset and AKI cessation during index hospitalization
Time Frame: Assessed from the point of randomization to the point of AKI cessation during index hospitalization, up to 365 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Usual Care | Drug-specific Alert
Number analyzed (Participants) | 2528 | 2532
days | 1.1 [0.8 to 2.2] | 1 [0.8 to 2.1]

11. Secondary Outcome: Readmission Rate
Description: Number of readmissions within 30 days of discharge from index hospitalization
Time Frame: Within 30 days of index hospitalization discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Drug-specific Alert
Number analyzed (Participants) | 2528 | 2532
Participants | 354 | 322

12. Secondary Outcome: Index Hospitalization Cost
Description: Total cost of index hospitalization
Time Frame: Assessed from point of randomization to the date of discharge from index hospitalization, up to 365 days post randomization
Measure: Median (Inter-Quartile Range); unit: dollars
Arm/Group | Usual Care | Drug-specific Alert
Number analyzed (Participants) | 2528 | 2532
dollars | 27900 [12500 to 63400] | 26900 [12400 to 63600]

13. Secondary Outcome: Percentage of AKI "Best Practices" Achieved Per Subject During Index Hospitalization
Description: Best practices assessed include: Avoidance of nephrotoxins (cessation of order or absence of de novo order of IV constrast agent, aminoglycoside, NSAID, or ACE inhibitor within 24 hours of randomization), fluid administration (administration of fluids within 24 hours of randomization), urinalysis order (with or without microscopy within 24 hours of randomization), documentation of AKI (by ICD-9 and ICD-10 codes during index hospitalization), monitoring of creatinine (at least one serum creatinine measurement occurring within 36 hours of randomization), documentation of urine output (within 24 hours of randomization), renal consult order during index hospitalization.
  Each metric above is binary. Outcome is reported as a composite best practice outcome representing the proportion of best practices achieved per subject.
Time Frame: Assessed from 24 hours from randomization up to discharge of index hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Drug-specific Alert
Number analyzed (Participants) | 2528 | 2532
Participants
  Contrast administration | 502 | 519
  Fluid administration | 1572 | 1537
  Aminoglycoside administration | 20 | 18
  NSAID administration | 264 | 245
  ACEi administration | 377 | 316
  Urinalysis order | 1013 | 1024
  Documentation of AKI | 956 | 1000
  Monitoring of creatinine | 2325 | 2331
  Monitoring of urine output | 2085 | 2104
  Renal consult | 392 | 393

14. Secondary Outcome: Percentage of Subjects With Chart Documentation of AKI
Description: Percentage of subjects with chart documentation of AKI by post-discharge ICD-10 codes and by chart adjudication
Time Frame: Assessed from time of randomization through to date of index hospitalization discharge, up to 365 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Drug-specific Alert
Number analyzed (Participants) | 2528 | 2532
Participants | 956 | 1000

ADVERSE EVENTS:
Time Frame: From randomization to index hospital discharge, up to 365 days
Description: An adverse event would require a temporary or permanent interruption of study activities and would be reported to the IRB within 5 calendar days of the Principal Investigator becoming aware of the event.
Arm/Group | Usual Care | Drug-specific Alert
All-Cause Mortality (participants affected / at risk) | 365/2528 | 356/2532
Serious Adverse Events (participants affected / at risk) | 0/2528 | 0/2532
Other Adverse Events (participants affected / at risk) | 0/2528 | 0/2532

LIMITATIONS AND CAVEATS:
Limitations include the fact that only three medication classes were targeted, that this trial was randomized at the patient level, which introduces the possibility of contamination, that it was conducted within a single health system, potentially limiting generalizability, that alert fatigue may have diminished alert performance as it was displayed in competition with all other alerts, and that the language of the alert was limited in how stringently it could recommend medication cessation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT02771977/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT02771977/ICF_001.pdf